CLINICAL TRIAL: NCT01033331
Title: Evaluation of the Muscle Strength and Motor Ability in Children With Spinal Muscle Atrophy Type II and III Treated With Valproic Acid
Brief Title: Evaluation of the Muscle Strength and Motor Ability in Children With Spinal Muscle Atrophy(SMA) Treated With Valproic Acid
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Evaluation of the muscle strength and motor ability in type II and III spinal muscle atrophy children treated with valproic acid, University of Sao PAulo General Hospital
Other Study IDs: 290/06; CAPES9030 (Other Grant/Funding Number: CAPES)
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2009-12-16 (Estimated); Status verified 2008-08

CONDITIONS: Spinal Muscular Atrophy
Keywords: Spinal Muscular atrophy; Valproic acid; HMAS; MRC scale
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if the treatment with valproic acid can increase the muscle strength and motor ability of children with spinal muscular atrophy.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is an autosomal recessive disorder that affects the motoneurons of the spinal anterior corn, resulting in hypotonia and muscle weakness. The knowledge about its molecular mechanism has led to clinical tests with drugs that increase survival motor neuron (SMN) protein level. The valproic acid (VA) that acts as a histone deacetylase inhibitor activates the SMN2 gene increasing the protein level. Methods: Twenty-two patients with type II and III SMA, aged between 2 and 18 years old, were treated with VA and were evaluated five times along a period of one year using the Manual Muscle Test (Medical Research Council scale-MRC), the Hammersmith Motor Ability Score, and the Barthel Index. The first evaluation was coincident with the introduction of VA. Results: After 12 months of therapy, the patients did not gain muscle strength but their motor ability has improved. Children younger than 6 years of age had a higher pronounced gain in motor ability. Conclusion: treatment of SMA patients with VA is one alternative to alleviate the progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Regularly attended at the Out-patient Service of Neuromuscular Disorders and Child Neurology of our Institution;
* More than 2 years olf and had a molecular analysis of Spinal Muscular Atrophy;

Exclusion Criteria:

* Had been submitted into a surgery recently;
* Did not come to the evaluation and medical sessions:
* Did not take the medication correctly

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 22 children with spinal muscular atrophy disease
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Test (Medical Research Council scale-MRC), the Hammersmith Motor Ability Score | one year

SECONDARY OUTCOMES:
Barthel Index | one year

CONTACTS AND LOCATIONS:
Overall Officials: Umbertina Reed, Doctor, Principal Investigator — Sao Paulo University
Locations (1):
- Section of Neuromuscular Disorders and Service of Child Neurology, Clinics Hospital of the School of Medicine at São Paulo University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Swoboda KJ, Scott CB, Reyna SP, Prior TW, LaSalle B, Sorenson SL, Wood J, Acsadi G, Crawford TO, Kissel JT, Krosschell KJ, D'Anjou G, Bromberg MB, Schroth MK, Chan GM, Elsheikh B, Simard LR. Phase II open label study of valproic acid in spinal muscular atrophy. PLoS One. 2009;4(5):e5268. doi: 10.1371/journal.pone.0005268. Epub 2009 May 14. PMID 19440247
- [Derived] Darbar IA, Plaggert PG, Resende MB, Zanoteli E, Reed UC. Evaluation of muscle strength and motor abilities in children with type II and III spinal muscle atrophy treated with valproic acid. BMC Neurol. 2011 Mar 24;11:36. doi: 10.1186/1471-2377-11-36. PMID 21435220